CLINICAL TRIAL: NCT06464146
Title: Pain Reduction for Limb Injuries in Pediatric Emergency Departments: A Randomised Clinical Trial Comparing Intranasal Fentanyl or Intranasal Ketamine to Oral Morphine
Brief Title: Pain Reduction for Limb Injuries in Pediatric Emergency Departments: Intranasal Fentanyl or Intranasal Ketamine vs Oral Morphine
Acronym: ANTAMIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP211044; 2023-506803-25 (EudraCT Number)
Record Dates: First submitted 2024-06-03; First posted 2024-06-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Limb Injury
Keywords: Fentanyl; Ketamin; Limb injury; Pain; Children
MeSH Terms: conditions — Pain | interventions — Morphine; Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Morphine (Active Comparator): Oral morphine (0.5mg/kg) and IN placebo
  Interventions: Drug: Morphine; Drug: NaCl 0,9 %
- IN Fentanyl (Experimental): placebo of oral morphine and IN fentanyl (1.5 µg/kg)
  Interventions: Drug: IN fentanyl; Drug: NaCl 0,9 %
- IN Ketamin (Experimental): placebo of oral morphine and IN ketamine (1 mg/kg)
  Interventions: Drug: IN ketamine; Drug: NaCl 0,9 %

INTERVENTIONS:
Drug: Morphine — oral morphine (0.5 mg / kg)
  Arms: Morphine
Drug: IN fentanyl — IN fentanyl (1.5 µg/kg)
  Arms: IN Fentanyl
Drug: IN ketamine — IN ketamine (1 mg/kg)
  Arms: IN Ketamin
Drug: NaCl 0,9 % — Injectable solution used as Placebo of Oral morphine or IN fentanyl/ ketamine.

SUMMARY:
The purpose of this study is to determine if IN fentanyl (1.5 µg/kg) or IN ketamine (1 mg/kg) is more effective at 30 minutes than oral morphine (0.5 mg/kg) in reduction of moderate and severe pain associated with limb injuries in patients 2-17 years of age presenting to the ED.

DETAILED DESCRIPTION:
In children with moderate to severe pain due to musculoskeletal injuries, the first-line analgesic therapy in pediatric emergency departments (ED) is oral or intravenous morphine. Due to the delay or discomfort associated with establishing IV access, oral forms are preferred in French ED. Unfortunately, oral morphine alone or with ibuprofen or paracetamol, none regimen is optimal for relieving pain in children with traumatic limb injuries. However, the use of intranasal course is a safe route that can provide rapid and almost immediate analgesia. Intranasal administration is easy, non-invasive and usually well tolerated by children. In the last years, drugs with analgesic and sedative properties is increasing, particularly on fentanyl, ketamine, which can be also administered by the IN route. There are currently no studies, neither published nor ongoing, which compare IN fentanyl or IN ketamine to a standard oral morphine for children with acute moderate to severe pain with limb injuries presenting to the ED. The main hypothesis is that the efficacy of the analgesia 30 minutes after the administration will be higher with IN Fentanyl or with IN Ketamine, when compared to oral morphine.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 2 years to 17 years and 11 months
* With 10 kg ≤ Weight ≤ 100 kg
* Presenting to ED with a traumatic pain and suspected fracture(s) based on an acute deformity AND experiencing pain and/or functional impotence in the injured limb(s)
* Within the first 12 hours after the injury
* VAS pain score at ED arrival ≥ 60/100 (if child ≥ 7 years) or Evendol pain score at ED arrival ≥ 7/15 (if child < 7 years)
* Affiliated to health insurance
* At least one signed parental informed consent

Exclusion Criteria:

* Received narcotic pain medication prior to arrival
* Contraindication to morphine, mentioned in SmPC
* Hypersensitivity to ketamine or fentanyl or to excipients (sodium chloride, sodium hydroxide), or to other opioids.
* Contraindication to fentanyl or ketamine, mentioned in SmPC
* GCS <15
* Evidence of significant femur, head, chest, abdominal, or spine injury
* Open fracture
* Nasal trauma or complete nasal obstruction
* Active epistaxis
* Nasal or sinus surgery within 6 months before inclusion
* History of high blood pressure, known coronary artery disease, congestive heart failure, acute glaucoma, increased intracranial pressure, major psychiatric disorder, hepatocellular insufficiency
* Active or history of psychiatric disorder
* Known pregnancy or suspicion of being pregnant
* Breastfeeding
* Non-French speaking parent and / or child.
* Participation to another interventional clinical research

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Degree of pain (M30) | 30 minutes
  Success: children <7 years with a pain score assessed by Evendol < 5 years, 30 minutes after drugs administration, without rescue analgesia. Scale: 0-15 (no pain - painful)
Degree of pain (M30) | 30 minutes
  Success: children ≥ 7 years with pain score assessed by VAS ≤ 30, 30 minutes after drugs administration, without rescue analgesia. Visual Analog Scale : 0-100 (no pain- painful)

SECONDARY OUTCOMES:
Degree of pain (M15) | 15 minutes
  Success: children <7 years with a pain score assessed by Evendol < 5, 15 minutes after drugs administration, without rescue analgesia
Degree of pain (M15) | 15 minutes
  Success: children ≥ 7 years with pain score assessed by VAS ≤ 30, 15 minutes after drugs administration, without rescue analgesia
Degree of pain (M60) | 60 minutes
  Success: children <7 years with a pain score assessed by Evendol < 5, 60 minutes after drugs administration, without rescue analgesia
Degree of pain (M60) | 60 minutes
  Success: children ≥ 7 years with pain score assessed by VAS ≤ 30, 60 minutes after drugs administration, without rescue analgesia
Degree of pain (M90) | 90 minutes
  Success: children <7 years with a pain score assessed by Evendol < 5, 90 minutes after drugs administration, without rescue analgesia
Degree of pain (M90) | 90 minutes
  Success: children ≥ 7 years with pain score assessed by VAS ≤ 30, 90 minutes after drugs administration, without rescue analgesia
Degree of pain (M120) | 120 minutes
  Success: children <7 years with a pain score assessed by Evendol < 5, 120 minutes after drugs administration, without rescue analgesia
Degree of pain (M120) | 120 minutes
  Success: children ≥ 7 years with pain score assessed by VAS ≤ 30, 120 minutes after drugs administration, without rescue analgesia
Reduction in pain (M15) | 15 minutes
  Reduction in pain from baseline assessed by Evendol for children <7 years
Reduction in pain (M15) | 15 minutes
  Reduction in pain from baseline assessed by VAS for children ≥ 7 years
Reduction in pain (M30) | 30 minutes
  Reduction in pain from baseline assessed by Evendol for children <7 years
Reduction in pain (M30) | 30 minutes
  Reduction in pain from baseline assessed by VAS for children ≥ 7 years
Reduction in pain (M60) | 60 minutes
  Reduction in pain from baseline assessed by Evendol for children <7 years
Reduction in pain (M60) | 60 minutes
  Reduction in pain from baseline assessed by VAS for children ≥ 7 years
Reduction in pain (M90) | 90 minutes
  Reduction in pain from baseline (assessed by VAS for children ≥ 7 years)
Reduction in pain (M90) | 90 minutes
  Reduction in pain from baseline assessed by Evendol for children <7 years
Reduction in pain (M120) | 120 minutes
  Reduction in pain from baseline assessed by VAS for children ≥ 7 years
Reduction in pain (M120) | 120 minutes
  Reduction in pain from baseline assessed by EVENDOL for children < 7 years
Degree of pain (M30) for comparison ketamine vs fentanyl | 30 minutes
  Success pain evaluation, as defined in primary outcome (for the comparison between ketamine and fentanyl) assessed by Evendol for children <7 years
Degree of pain (M30) for comparison ketamine vs fentanyl | 30 minutes
  Success pain evaluation, as defined in primary outcome (for the comparison between ketamine and fentanyl) assessed by VAS for children ≥ 7 years
Level of sedation (M5) | 5 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Level of sedation (M10) | 10 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Level of sedation (M15) | 15 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Level of sedation (M30) | 30 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Level of sedation (M60) | 60 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Level of sedation (M90) | 90 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Level of sedation (M120) | 120 minutes
  Level of sedation as measured by the University of Michigan Sedation Scale Score (UMSS) after drugs administration, from 0 (patient awake) to 4 (patient unawakable)
Number of participants with Adverse events | From study treatment intake until ED discharge, up to 1 day
  Adverse events potentially associated with IN ketamine, IN fentanyl and/or oral morphine: drowsiness, dizziness, pruritus, nausea, vomiting, dysphoria, nasal burning and irritation, unpleasant taste, vision changes, throat irritation, headache, vital sign changes (heart rate, respiratory rate, oxygen saturation, blood pressure).
Score of satisfaction | At ED discharge, up to 1 day
  General satisfaction of parents and patient ≥ 7 years old on a scale of 0-100 with corresponding faces (0 = no satisfaction at all, 100 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène CHAPPUY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Roger Salengro Hospital, Lille
  - Timone Hospital, Marseille
  - Mère-Enfant Hospital, Nantes
  - Hopital Necker Enfants malades, Paris

IPD SHARING:
Plan to Share IPD: No